CLINICAL TRIAL: NCT03875443
Title: Structured Educational Program and the Use of a Practical Algorithm for Reduction and Stabilisation of Trochanteric Fractures With in Intramedullary Nail Improved Radiologic Reduction and Implant Positioning. A Prospective Study With 6 Months Follow-up.
Brief Title: Trochanteric Fractures - How to Improve the Results of Reduction and Implant Positioning
Acronym: PERTROCH
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00025; ch19Eckardt
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Hip Fractures
Keywords: implant positioning; reduction; intraoperative fluoroscopy; reduction algorithm
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Instructional video — Video (produced by AO Trauma and Prof. Daniel Rikli) includes a stepwise and structured explanation of the different fluoroscopic views necessary to evaluate intraoperatively with the fluoroscope different aspects of the proximal femur. The video is publically available under: (https://www.aointeract.org/#/watch/video/L3YxL3ZpZGVvcy8xOTc=/intraoperative-imaging-of-femur).
Other: Reduction algorithm — Intraoperative reduction algorithm (developed by PD Henrik Eckardt); each step in the algorithm will be checked and documented with the fluoroscope and archived using the store function of the fluoroscope.

SUMMARY:
This prospective study (including patients with an intertrochanteric or subtrochanteric fractures type 31A1, 31A2 and 31A3) is to assess the effect of an educational intervention for operating surgeons with respect to an improvement of the quality of reduction and internal stabilisation of intertrochanteric fractures. A historic cohort of patients operated at the University Hospital Basel for an intertrochanteric fracture from 2014-2015 will be used for comparison.

DETAILED DESCRIPTION:
Intertrochanteric fractures are one of the most frequent fracture type in the elderly population usually occurring in patients older than 60 years of age. Almost all fractures are treated operatively with reduction and stabilisation of the fracture using either a dynamic hip screw or an intramedullary nail. The reduction of the fracture and positioning of the implant are surgeon dependent factors and can be influenced by educational interventions. The investigators hypothesized that a structured educational program on the optimal use of intraoperative fluoroscopy to control the quality of reduction and the position of the implant, as well as the provision of a practical algorithm intraoperatively guiding reduction and stabilisation of intertrochanteric fractures would improve the radiologic outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with an intertrochanteric fracture type 31A1 or 31A2 or subtrochanteric fracture type 31A3
* Surgeon must have completed the teaching video on how to evaluate intraoperatively the fracture, the reduction and the implant positioning and complete the reduction algorithm documenting that all intraoperative steps have been correctly accomplished

Exclusion Criteria:

* Patients operated without adherence to the reduction algorithm
* Patients operated by surgeons who did not attend the teaching session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with an intertrochanteric fracture or subtrochanteric fracture at the Department of Orthopaedic and Traumatology, University Hospital Basel
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Shortening of the femoral neck (mm) | 6 months after hip surgery
  Radiologic result: Shortening of the femoral neck as measured with sliding of the femoral neck screw inside the nail
Change of the shaft-neck angle (degree) | 6 months after hip surgery
  Radiologic result: Change of the shaft-neck angle on the antero-posterior view in comparison to postoperative value
Displacement of the calcar segment in the lateral view | 6 months after hip surgery
  Radiologic result: Displacement of the calcar segment in the lateral view
Central placement of the femoral neck screw (degree) | 6 months after hip surgery
  Radiologic result: Central placement of the femoral neck screw as measured with the Tip-Apex-Distance

SECONDARY OUTCOMES:
Hip re-operations | 6 months after hip surgery
  Number of re-operations due to loss of reduction
Mortality | 6 months after hip surgery
  Number of patients that have died
Operation time from incision until closure of the wound (minutes) | second postoperative day
  Operation time from incision until closure of the wound
Central placement of the femoral neck screw (degree) | second postoperative day
  Radiologic result: Central placement of the femoral neck screw as measured with the Tip-Apex-Distance
Reduction of the calcar segment in the lateral view (mm) | second postoperative day
  Radiologic result: Reduction of the calcar segment in the lateral view

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Eckardt, PD Dr. med, Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland